CLINICAL TRIAL: NCT02730039
Title: Meaning-Centered Psychotherapy Training for Cancer Care Providers
Status: Active, not recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Stanford University (Other); Northwestern University (Other); MJHS Institute for Innovation in Palliative Care (Other); Massachusetts General Hospital (Other); City of Hope Medical Center (Other); Dana-Farber Cancer Institute (Other); New York Presbyterian Hospital (Other); Odette Cancer Center - Sunnybrook Hospital (Unknown); VA New York Harbor Healthcare System (U.S. Federal Agency); University of Pennsylvania (Other); Smilow Cancer Hospital - Yale New Haven Health (Unknown); Department of Veterans Affairs, New Jersey (U.S. Federal Agency); Vidant Cancer Care (Unknown)
Responsible Party: Sponsor
Other Study IDs: 15-321
Record Dates: First submitted 2016-03-15; First posted 2016-04-06 (Estimated); Last update posted 2025-12-30 (Actual); Status verified 2025-01

CONDITIONS: Cancer Care Providers
Keywords: Cancer Care Providers; Psychotherapy; 15-321

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cancer Care Providers: Provider will attend a MCPT two-day intensive workshop that will include:
  * Didactic Components
  * Experiential Exercises
  * Simulated patient role plays with actors
  * Provider completes MCPT Workshop Assessment MCPT POST-WORKSHOP IMPLEMTATION (OPTIONAL)
  * MCP Core Competency Trainer rated Assessment
  * MCP Pre & Post Workshop Knowledge Assessment
  * MCPT Session Evaluation Assessment Provider will participate in training follow-up calls & webinars for approximately 6 -12 months following completion of MCPT workshop.
  * Provider will have ongoing access to MCPT Website with a discussion board, training resources and materials for clinical care.
  * Provider will complete follow-up assessment at 3, 6, 9, & 12 months post-training
  * Training Update
  * Goal Evaluation Form
  * MCP Core Competency Self-Assessment MCPT POST-WORKSHOP IMPLEMTATION (OPTIONAL)
  Interventions: Behavioral: workshop; Behavioral: follow-up calls & webinars; Behavioral: assessments

INTERVENTIONS:
Behavioral: workshop
Behavioral: follow-up calls & webinars
Behavioral: assessments

SUMMARY:
The purpose of this project, entitled "Meaning-Centered Psychotherapy Training for Cancer Care Providers," is to develop a multi-modal training program in Meaning-Centered Psychotherapy (MCP) for multidisciplinary cancer care clinicians who provide psycho-oncology and psychosocial palliative care services for cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Clinicians who provide psycho-oncology and/or psychosocial palliative care services for to patients with cancer and/or severe medical illness/disease at MSKCC, other institutions, or in the community, as per self-report.
* Completed online MCPT application form and commits to attend the two-day intensive MCPT program, complete training follow-up assessments, and participate in required follow-up training activities.
* Able to speak, read, and understand English proficiently to participate in MCPT training sessions and complete assessments.

Exclusion Criteria:

* Does not meet the criteria of an appropriate candidate for training program, as determined by review of the MCPT Application Evaluation Checklist in the opinion of the investigator.

  * Materials for the training and the training will be conducted in English only.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: clinicians (20% MSKCC providers & 80% outside providers)
Sampling Method: Non-Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2015-12-11 (Actual); Primary Completion 2026-12-11 (Estimated); Study Completion 2026-12-11 (Estimated)

PRIMARY OUTCOMES:
participant's skills uptake at the end of the MCPT session score range 0-10 | change from Baseline to 12 months
  Evaluation will take place on two levels, as data will be collected directly from: 1) MCPT participants and 2) MCP trainers. Data on the training will be collected before and during the MCPT session. Data on post-MCP training will be collected for one year following participation in the MCPT.

CONTACTS AND LOCATIONS:
Overall Officials: William Breitbart, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/